CLINICAL TRIAL: NCT04544995
Title: A Phase 1, Multicentre, Open-Label, Dose-Escalation and Cohort Expansion Study of Niraparib and Dostarlimab in Paediatric Patients With Recurrent or Refractory Solid Tumours
Brief Title: Dose Escalation and Cohort Expansion Study of Niraparib and Dostarlimab in Paediatric Participants With Solid Tumors (SCOOP)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 213406; 2020-002359-39 (EudraCT Number)
Record Dates: First submitted 2020-09-04; First posted 2020-09-10 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
Keywords: Dose escalation; Dose expansion; Dostarlimab; Niraparib; Osteosarcoma; Neuroblastoma
MeSH Terms: conditions — Neoplasms; Osteosarcoma; Neuroblastoma | interventions — niraparib; Tablets; Suspensions; dostarlimab

STUDY DESIGN:
Masking Description: This will be an open-label study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Part 1A: Dose Escalation (Experimental): Participants with body weight of ≥ 20 kilogram (kg) and who can swallow niraparib tablets will receive niraparib tablets and dostarlimab.
  Interventions: Drug: Dostarlimab; Drug: Niraparib (Tablet)
- Part 1B: Dose Escalation (Experimental): Participants who are <8 years of age will receive niraparib TfOS and dostarlimab.
  Interventions: Drug: Niraparib (Tablet for oral suspension); Drug: Dostarlimab
- Part 2 Safety Run-in (Experimental): Participants with osteosarcoma or neuroblastoma who are ≥8 years of age will receive niraparib TfOS and dostarlimab.
  Interventions: Drug: Niraparib (Tablet for oral suspension); Drug: Dostarlimab
- Part 2A: Cohort Expansion for Osteosarcoma (Experimental): Participants with osteosarcoma will receive the RP2D of the combination of niraparib and dostarlimab.
  Interventions: Drug: Niraparib (Tablet for oral suspension); Drug: Dostarlimab; Drug: Niraparib (Tablet)
- Part 2B: Cohort Expansion for Neuroblastoma (Experimental): Participants with neuroblastoma will receive the RP2D of the combination of niraparib and dostarlimab.
  Interventions: Drug: Niraparib (Tablet for oral suspension); Drug: Dostarlimab; Drug: Niraparib (Tablet)

INTERVENTIONS:
Drug: Niraparib (Tablet for oral suspension) — Niraparib will be administered as TfOS (Tablet for oral suspension)
  Arms: Part 1B: Dose Escalation; Part 2 Safety Run-in; Part 2A: Cohort Expansion for Osteosarcoma; Part 2B: Cohort Expansion for Neuroblastoma
Drug: Dostarlimab — Dostarlimab will be administered as IV infusion
Drug: Niraparib (Tablet) — Niraparib will be administered as tablet
  Arms: Part 1A: Dose Escalation; Part 2A: Cohort Expansion for Osteosarcoma; Part 2B: Cohort Expansion for Neuroblastoma

SUMMARY:
This study will evaluate the combination of a poly (adenosine diphosphate-ribose) polymerase (PARP) inhibitor, niraparib, with the programmed cell death protein 1 (PD-1) inhibitor, dostarlimab in the paediatric population. This study will be conducted to determine the recommended Phase 2 dose (RP2D) and evaluate the pharmacokinetics (PK), safety, and efficacy of niraparib in combination with dostarlimab in paediatric participants with recurrent or refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

For Part 1 and Part 2:

* Participant is a child or an adolescent greater than or equal to (>=) 6 months to less than (<) 18 years old at the time of informed consent/assent.
* Participant with disease other than neuroblastoma has radiologically measurable disease at screening that can be tracked as RECIST v1.1 target lesion(s).
* Participant with neuroblastoma has measurable/evaluable target and/or non-target disease by INRC at screening. Neuroblastoma participants with recurrent/relapsed bone metastasis that is metaiodobenzylguanidine (MIBG)-positive (or FDG-PET positive, for MIBG-nonavid tumors) as only site of disease are eligible.
* Performance status must be >=60 percent on the Karnofsky scale for participants >16 years of age and >=60 percent on the Lansky scale for participants less than or equal to (<=) 16 years of age.
* Participant has adequate organ function.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP) or Is a WOCBP and using a contraceptive method that is highly effective.
* A male participant of reproductive potential is eligible to participate if he agrees to refrain from donating sperm plus, either be abstinent from heterosexual intercourse or must agree to use a male condom starting with the first dose of study treatment through at least 90 days after the last dose of study treatment.

For Part 1 only:

• Participant has recurrent or refractory osteosarcoma, neuroblastoma, adrenocortical carcinoma, Ewing sarcoma, rhabdomyosarcoma, or any other solid tumor (excluding tumors of the central nervous system [CNS]) and must not be eligible for alternative curative treatment: i. Participants with non-CNS solid tumours other than osteosarcoma, neuroblastoma, adrenocortical carcinoma, Ewing sarcoma or rhabdomyosarcoma are required to have prior documented breast cancer susceptibility gene (BRCAness) mutational signature (mutational signature 3) on deoxyribonucleic acid (DNA) sequencing of tumor obtained in the relapsed/recurrent disease setting, within 6 (preferably 3) months of Cycle 1 Day 1.

ii. For participants with documented BRCAness mutational signature: Existing information on molecular profiling of the participant's tumor tissue must be through a molecular profiling platform such as Individualized Therapy for Relapsed Malignancies in Childhood (INFORM). Molecular profile information must contain information from whole exome sequencing or whole genome sequencing, including the mutation status of BRCA1 and BRCA 2 and other homologous recombination DNA repair (HRR) pathway genes, mutational signatures including mutational signature 3, and tumor mutational burden (TMB).

iii. NOTE: Participants with recurrent or refractory osteosarcoma, neuroblastoma, adrenocortical carcinoma, Ewing sarcoma, or rhabdomyosarcoma are asked to provide documentation, if available, of the BRCAness mutational signature analysis on DNA sequencing of their tumour.

For Part 2A:

• Participant has recurrent or refractory osteosarcoma and must not be eligible for alternative curative treatment.

Documentation of BRCAness mutational signature 3 will be requested, but not required, for enrollment.

• Participant must confirm at screening that an archival or fresh tumor tissue sample is available for use, in retrospective exploratory biomarker analysis. Otherwise, enrolling site must discuss with Sponsor.

For Part 2B:

* Participant has recurrent or refractory neuroblastoma and must not be eligible for alternative curative treatment. Documentation of BRCAness mutational signature 3 will be requested, but not required, for enrollment.
* Participant must confirm at screening that an archival or fresh tumor tissue sample is available for use, in retrospective exploratory biomarker analysis. Otherwise, enrolling site must discuss with Sponsor.

Exclusion Criteria:

For Part 1 and Part 2:

* Participant has known hypersensitivity to dostarlimab or niraparib, their components, or their excipients.
* Participant has a known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* Participant has active autoimmune disease that has required systemic treatment in the past 2 years (that is [i.e.], with use of disease-modifying anti-rheumatic drugs, corticosteroids, or immunosuppressive drugs). Replacement therapy (for example [e.g.], thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Participant has known active CNS metastases, carcinomatous meningitis, or both. Carcinomatous meningitis precludes a participant from study participation regardless of clinical stability.
* Participant had a known additional (second primary) malignancy that progressed or required active treatment within the last 2 years.
* Participant is considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or active infection that requires systemic therapy.
* Participant has a condition (such as transfusion-dependent anemia or thrombocytopenia), requirement for therapy, or laboratory abnormality that might confound the study results or interfere with the participant's participation for the full duration of the study treatment.
* Participant has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Participant has a known history of human immunodeficiency virus (HIV) (type 1 or 2 antibodies).
* Participant has documented presence of HbsAg and/or HBcAb at Screening or within 3 months prior to first dose of study intervention. Participants with a negative HbsAg and positive HbcAb result are eligible only if HBV DNA is negative.
* Participant must not have a gastrointestinal condition, such as bowel obstruction, that can impact absorption of oral medications and is identified by clinical symptoms or CT scan, etc.
* Participant has had any known Grade 3 or 4 anemia, neutropenia, and/or thrombocytopenia that was related to the most recent prior anti-cancer treatment and that persisted >4 weeks (28 days).
* Participant has not recovered (i.e., to Grade ≤1 or to baseline) from prior systemic anticancer therapy-induced AEs. Note: Participants with alopecia, hearing impairment, Grade ≤2 neuropathy, Grade ≤2 fatigue, Grade ≤ 2 anaemia, and/or Grade ≤2 neutropenia are an exception to this criterion and may qualify for participation in the study.
* Participant had toxicity related to prior immunotherapy that led to study treatment discontinuation.
* Participant had treatment with systemic anticancer therapy (investigational agent or device, or approved chemotherapy, targeted therapy, immunotherapy, or other systemic therapy) within 3 weeks or 5 half-lives, whichever is shorter, prior to the first dose of study treatment, radiation therapy encompassing >20 percent of the bone marrow within 2 weeks prior to the first dose of study treatment, or any radiation therapy within 1 week prior to the first dose of study treatment.
* Participant has not recovered adequately from AEs or complications from any major surgery prior to starting study treatment.
* Participant has received a live vaccine within 30 days of planned start of study treatment.
* Participant has clinically significant cardiovascular disease (e.g., significant cardiac conduction abnormalities, uncontrolled hypertension, cardiac arrhythmia or unstable angina, New York Heart Association Grade 2 or greater congestive heart failure, serious cardiac arrhythmia requiring medication, and history of cerebrovascular accident) within 6 months of enrolment.
* Participant has heart rate-corrected QT interval prolongation at screening >450 milliseconds (msec) or >480 msec for participants with bundle branch block.
* Participant has received a solid organ transplant.
* Participant has a documented presence of HCV antibody at Screening or within 3 months prior to first dose of study intervention. NOTE: Participants with a positive HCV antibody test result due to prior resolved disease can be enrolled, if a confirmatory HCV RNA test is negative and the participant otherwise meets entry criteria.
* Participant has a documented presence of HCV RNA at Screening or within 3 months prior to first dose of study intervention. NOTE: The HCV RNA test is optional and participants with negative HCV antibody test are not required to undergo HCV RNA testing as well.

For Part 2:

* Participant has received prior therapy with an anti-PD-1, anti-programmed cell death ligand 1, anti-programmed cell death-ligand 2, anti-cytotoxic T-lymphocyte-associated antigen-4 antibody (including ipilimumab), or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways (with the exception of participants rolling over from Part 1 of the study: these participants are allowed to have received dostarlimab).
* Participant has had prior treatment with a known poly(adenosine diphosphate-ribose) polymerase (PARP) inhibitor (with the exception of participants rolling over from Part 1 of the study: these participants are allowed to have received niraparib).

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was performed in two parts: Part 1: Dose Escalation and Part 2: Safety Run-in and Cohort Expansion.
Groups:
- Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg): Paediatric participants with recurrent or refractory solid tumours received 100 mg niraparib tablet orally once daily along with 3 mg/kg dostarlimab solution as a 30-minute intravenous (IV) infusion prior to the niraparib dose on Day 1 of each 21-day treatment cycle until the end of treatment period, disease progression (PD), unacceptable toxicity, withdrawal of consent/assent, investigator's decision to withdraw, or death.
- Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg: Paediatric participants with recurrent or refractory solid tumours received 100 mg niraparib tablet orally once daily along with 7.5 mg/kg dostarlimab solution as a 30-minute IV infusion prior to the niraparib dose on Day 1 of each 21-day treatment cycle until the end of treatment period, PD, unacceptable toxicity, withdrawal of consent/assent, investigator's decision to withdraw, or death.
- Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg: Paediatric participants with recurrent or refractory solid tumours received 200 mg niraparib tablet orally once daily along with 3 mg/kg dostarlimab solution as a 30-minute IV infusion prior to the niraparib dose on Day 1 of each 21-day treatment cycle until the end of treatment period, PD, unacceptable toxicity, withdrawal of consent/assent, investigator's decision to withdraw, or death.
- Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg: Paediatric participants with recurrent or refractory solid tumours received niraparib (age-based dose) age-appropriate liquid formulation (AAOLF) orally once daily and 7.5 mg/kg dostarlimab as a 30-minute IV infusion before the niraparib dose on Day 1 of each 21-day cycle until the end of the Treatment Period, PD, unacceptable toxicity, withdrawal of consent/assent, investigator's decision, or death.
- Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma): Paediatric participants with recurrent or refractory osteosarcoma received 100 mg niraparib tablet orally once daily along with 7.5 mg/kg dostarlimab solution as a 30-minute intravenous (IV) infusion prior to the niraparib dose on Day 1 of each 21-day treatment cycle until the end of treatment period, PD, unacceptable toxicity, withdrawal of consent/assent, investigator's decision to withdraw, or death.
- Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma): Paediatric participants with recurrent or refractory neuroblastoma received 100 mg niraparib tablet orally once daily along with 7.5 mg/kg dostarlimab solution as a 30-minute intravenous (IV) infusion prior to the niraparib dose on Day 1 of each 21-day treatment cycle until the end of treatment period, PD, unacceptable toxicity, withdrawal of consent/assent, investigator's decision to withdraw, or death.
- Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg: Paediatric participants with recurrent or refractory osteosarcoma or neuroblastoma received niraparib (dose based on weight) tablet for oral suspension (TfOS) orally once daily along with 7.5 mg/kg dostarlimab solution as a 30-minute intravenous (IV) infusion prior to the niraparib dose on Day 1 of each 21-day treatment cycle until the end of treatment period, PD, unacceptable toxicity, withdrawal of consent/assent, investigator's decision to withdraw, or death.
Period: Overall Study
Arm/Group | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma) | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma) | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg
Started (The safety population is defined as all participants who received at least 1 dose of either niraparib or dostarlimab.) | 11 | 7 | 5 | 3 | 11 | 7 | 3
DLT-Evaluable Population (The DLT-evaluable population included participants from Part 1 or Part 2 Safety Run-in who completed the DLT observation period through at least 2 cycles of study treatment (including ≥80% of the intended niraparib dose and ≥2 infusions of dostarlimab) or experienced a DLT. For the thrombocytopenia event endpoint, participants were included if they experienced Grade ≥3 thrombocytopenia adverse events during the observation period) | 8 | 6 | 2 | 2 | 0 | 0 | 3
Intent-to-Treat (ITT) Population (The ITT population included all participants who received any study medication and had measurable baseline tumour assessment.) | 11 | 6 | 5 | 3 | 0 | 0 | 3
Modified Intent-to-Treat (mITT) Population (The mITT Population included all participants who received any study medication, had measurable baseline tumour assessment, and/or, for neuroblastoma participants, MIBG-positive disease (or FDG-positive disease, for MIBG-nonavidtumours) at baseline, and had at least 1 postbaseline tumour assessment) | 0 | 0 | 0 | 0 | 9 (1 participant treated in Part 1A Cohort 1A is mITT eligible and analyzed in this cohort.) | 8 (2 participants treated in Part 1A Cohort 1A are mITT eligible and analyzed in this cohort.) | 0
Pharmacokinetic (PK) Population (The PK population included all participants who received any amount of study drug and have ≥1 PK sample.) | 11 | 7 | 5 | 3 | 11 | 7 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 11 | 7 | 5 | 3 | 11 | 7 | 3
Not completed — Death | 7 | 3 | 3 | 3 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Reached protocol-defined stopping criteria | 3 | 4 | 2 | 0 | 4 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg: Paediatric participants with recurrent or refractory solid tumours received niraparib (dose based on age) age-appropriate liquid formulation (AAOLF) orally once daily and 7.5 mg/kg dostarlimab as a 30-minute IV infusion before the niraparib dose on Day 1 of each 21-day cycle until the end of the Treatment Period, PD, unacceptable toxicity, withdrawal of consent/assent, investigator's decision, or death.
- Total: Total of all reporting groups
Arm/Group | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma) | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma) | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg | Total
Number analyzed (Participants) | 11 | 7 | 5 | 3 | 11 | 7 | 3 | 47
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 13.9 (2.84) | 13.7 (3.99) | 13.0 (3.81) | 6.0 (1.00) | 14.3 (2.45) | 10.1 (2.97) | 14.7 (1.53) | 12.9 (3.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 3 | 3 | 5 | 3 | 2 | 22
  Male | 10 | 2 | 2 | 0 | 6 | 4 | 1 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 11 | 7 | 5 | 3 | 9 | 5 | 3 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1A and Part 1B: Number of Participants With Dose-limiting Toxicities (DLT)
Description: DLT referred to adverse effects within the first 42 days of treatment, indicating the maximum tolerated dose. DLTs included treatment-related Grade (G) 4 non-haematologic AEs or G3 AEs unresolved to G≤1 within 48 hours. G3/4 non-haematologic lab abnormalities were DLTs if causing hospitalization or persisting ≥7 days with symptoms or requiring intervention. Haematologic DLTs included prolonged G4 thrombocytopenia, G3/4 thrombocytopenia with bleeding or transfusion needs, prolonged G4 neutropenia, G3/4 neutropenia with infection, and G3/4 anemia requiring transfusion. Other criteria included Cycle 2 delays >2 weeks, unresolved G≥2 uveitis/endocrine toxicity, persistent colitis/diarrhea, unresolved G3/4 immune-related AEs, G≥3 infusion reactions, hemophagocytic lymphohistiocytosis, posterior reversible encephalopathy syndrome, and treatment-related G5 AE. DLT-evaluable participants completed ≥2 cycles with ≥80% of planned niraparib and ≥2 dostarlimab infusions or had a DLT.
Time Frame: Up to 42 days
Population: DLT-evaluable population consists of participants in Part 1 who completed the DLT observation period through at least 2 cycles of study treatment (including ≥80% of the intended niraparib dose and ≥2 infusions of dostarlimab) or experienced a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 8 | 6 | 2 | 2
Participants | 1 | 1 | 2 | 2

2. Primary Outcome: Part 2 Safety-run in: Number of Participants With Dose-limiting Toxicities (DLT)
Description: as for outcome 1
Time Frame: Up to 42 days
Population: DLT-evaluable Population consists of participants in Part 2 Safety Run-in who completed the DLT observation period through at least 2 cycles of study treatment (including ≥80% of the intended niraparib dose and ≥2 infusions of dostarlimab) or experienced a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 3
Participants | 1

3. Primary Outcome: Part 2 Safety-run in: Number of Participants With Grade ≥3 Thrombocytopenia Adverse Events
Description: Thrombocytopenia events were defined as treatment-related toxicities of Grade 3 or Grade 4 thrombocytopenia occurring within the first 42 days of study treatment. AEs were graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0.
Time Frame: Up to 42 days
Population: DLT-evaluable Population consists of participants in Part 2 Safety Run-in who completed the DLT observation period through at least 2 cycles of study treatment (including ≥80% of the intended niraparib dose and ≥2 infusions of dostarlimab) or experienced Grade ≥3 thrombocytopenia AEs.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Safety- Run-In Niraparib TfOS (Weight- Based Dose) + Dostarlima b 7.5 mg/kg: Paediatric participants with recurrent or refractory osteosarcoma or neuroblastoma received niraparib (dose based on weight) tablet for oral suspension (TfOS) orally once daily along with 7.5 mg/kg dostarlimab solution as a 30-minute intravenous (IV) infusion prior to the niraparib dose on Day 1 of each 21-day treatment cycle until the end of treatment period, PD, unacceptable toxicity, withdrawal of consent/assent, investigator's decision to withdraw, or death.
Arm/Group | Part 2: Safety- Run-In Niraparib TfOS (Weight- Based Dose) + Dostarlima b 7.5 mg/kg
Number analyzed (Participants) | 3
Participants | 0

4. Primary Outcome: Part 2A: Progression-Free Survival at 6 Months Per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1
Description: PFS6 is defined as the percentage of participants without progressive disease (PD) per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 or death at 6 months from the date of the first dose of study treatment. PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start).
Time Frame: At Month 6
Population: Modified Intent-to-treat (mITT) population for Part 2A Osteosarcoma cohort included participants who received any study medication, had measurable baseline tumour assessment, and had at least 1 post-baseline tumour assessment. Data from 1 participant treated in Part 1A Cohort 1A at the same dose level as 8 participants treated in Part 2A were pooled and analyzed collectively for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma)
Number analyzed (Participants) | 9
Percentage of Participants | 0 [0.0 to 33.6]

5. Primary Outcome: Part 2B: Objective Response Rate (ORR) by the Investigator Using International Neuroblastoma Response Criteria (INRC)
Description: ORR is defined as the percentage of participants who have a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) as determined by the Investigator using International Neuroblastoma Response Criteria (INRC). CR is resolution of all detectable disease, including soft tissue, bone, and bone marrow, with residual lesion measurements <10 mm and no tumor infiltration in the bone marrow or abnormal MIBG/FDG uptake. PR: Significant reduction in tumor burden, including a ≥30% decrease in primary or metastatic lesion size and ≥50% reduction in bone involvement (MIBG/FDG), with no new lesions and bone marrow infiltration ≤5%.
Time Frame: Up to approximately 196 weeks
Population: Modified Intent-to-treat (mITT) population for Part 2B Neuroblastoma cohort included participants who received any study medication, had measurable baseline tumour assessment and/or MIBG-positive disease (or FDG-positive disease, for MIBG-nonavid tumours) at baseline, and had at least 1 post-baseline tumour assessment. Data from 2 participants treated in Part 1A Cohort 1A at the same dose level as 6 participants treated in Part 2B were pooled and analyzed collectively for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma)
Number analyzed (Participants) | 8
Percentage of Participants | 0 [0.0 to 36.9]

6. Secondary Outcome: Part 1A and Part 1B: Objective Response Rate (ORR)
Description: ORR is the percentage of participants with a best overall response (BOR) of confirmed CR or PR using RECIST v1.1 or INRC (for neuroblastoma participants only) as determined by the Investigator. Per RECIST v1.1: CR is disappearance of all target lesions, with pathological lymph nodes <10 mm in short axis. PR is ≥30% decrease in sum of diameters of target lesions, referencing baseline sum (percent change from baseline). Per INRC: CR is resolution of all detectable disease, including soft tissue, bone, and bone marrow, with residual lesion measurements <10 mm and no tumor infiltration in the bone marrow or abnormal MIBG/FDG uptake. PR: Significant reduction in tumor burden, including a ≥30% decrease in primary or metastatic lesion size and ≥50% reduction in bone involvement (MIBG/FDG), with no new lesions and bone marrow infiltration ≤5%.
Time Frame: Up to approximately 196 weeks
Population: ITT Population included all participants who received any study medication and had measurable baseline tumour assessment and/or, for neuroblastoma participants, MIBG-positive disease (or FDG-positive disease, for MIBG-nonavid tumours) at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 11 | 6 | 5 | 3
Percentage of Participants | 9 [0.2 to 41.3] | 0 [0.0 to 45.9] | 0 [0.0 to 52.2] | 0 [0.0 to 70.8]

7. Secondary Outcome: Part 1A and Part 1B: Duration of Response (DOR)
Description: DOR is the time from first documented response (CR or PR) to first PD by RECIST v1.1 or INRC (neuroblastoma only), based on Investigator assessment, or death (whichever occurs first). If no PD or death occurs post-response, participants are censored at their last tumor assessment date. Per RECIST v1.1, CR is disappearance of all target lesions; PR is ≥30% decrease in lesion diameters from baseline; PD is ≥20% increase in lesion sum from nadir plus ≥5 mm absolute increase. Per INRC, CR is resolution of detectable disease, including soft tissue, bone, and bone marrow, with residual lesions <10 mm, no bone marrow infiltration, and normal MIBG/FDG uptake. PR is a ≥30% decrease in lesion size, ≥50% reduction in bone involvement (MIBG/FDG), no new lesions, and bone marrow infiltration ≤5%. PD is >20% lesion size increase, new lesions, or increased infiltration in bone marrow.
Time Frame: Up to approximately 196 weeks
Population: ITT population. Only responders (CR or PR) by investigator assessment were included in this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 1 | 0 | 0 | 0
Months | 37.29 [NA to NA] — Full range is not applicable as only a single participant was analyzed. |  |  |

8. Secondary Outcome: Part 1A and Part 1B: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A TEAE is any event that emerged during treatment and was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment. SAE is defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, or is a congenital anomaly/birth defect, other situations which involved medical or scientific judgment or is associated with liver injury and impaired liver function. SAEs are subset of AEs. AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA dictionary).
Time Frame: Up to approximately 196 weeks
Population: Safety Population is defined as all participants who received at least 1 dose of either niraparib or dostarlimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 11 | 7 | 5 | 3
Participants
  TEAEs | 11 | 7 | 5 | 3
  SAEs | 6 | 2 | 2 | 2

9. Secondary Outcome: Part 1A and Part 1B: Number of Participants With Dostarlimab-Related Immune-Mediated Adverse Events (imAEs)
Description: Dostarlimab-Related Immune-Mediated AEs were reported. AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA dictionary).
Time Frame: Up to approximately 196 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 11 | 7 | 5 | 3
Participants | 2 | 5 | 0 | 2

10. Secondary Outcome: Part 1A and Part 1B: Number of Participants With TEAEs Leading to Death and Treatment Discontinuation
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A TEAE is any event that emerged during treatment and was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment.
Time Frame: Up to approximately 196 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 11 | 7 | 5 | 3
Participants
  TEAEs leading to Death | 3 | 1 | 0 | 0
  Treatment Discontinuation | 3 | 1 | 1 | 2

11. Secondary Outcome: Part 1A and Part 1B: Niraparib Concentrations
Description: Blood samples were obtained to analyze niraparib concentration levels.
Time Frame: 2.5 hours (HR) and 7 HR post-dose on Cycle 1 Week 1, 168 HR post-dose on Cycle 1 Week 2
Population: Pharmacokinetic (PK) population included all participants who received at least one dose of study treatment and had at least one PK sample. Only those participants with data available at specified data points have been analyzed.
Measure: Mean (Standard Deviation); unit: nanogram/ millilitre (ng/mL)
Arm/Group | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 11 | 7 | 5 | 3
nanogram/ millilitre (ng/mL)
  Cycle 1 Week 1, 2.5 HR post-dose: number analyzed (Participants) | 11 | 7 | 5 | 2
  Cycle 1 Week 1, 2.5 HR post-dose | 120.045 (198.6774) | 44.300 (58.0753) | 83.480 (107.4614) | 383.900 (413.0918)
  Cycle 1 Week 1, 7 HR post-dose: number analyzed (Participants) | 9 | 7 | 5 | 2
  Cycle 1 Week 1, 7 HR post-dose | 347.889 (133.9846) | 254.571 (141.7096) | 640.200 (449.5850) | 522.500 (369.8168)
  Cycle 1 Week 2, 168 HR post-dose | 419.255 (203.6362) | 396.286 (276.8006) | 812.000 (704.5534) | 887.667 (628.3664)

12. Secondary Outcome: Part 1A and Part 1B: Dostarlimab Concentrations
Description: Blood samples were collected for PK analysis of Dostarlimab.
Time Frame: Pre-dose on Day 1; 1 HR post-dose on Cycle 1 Week 1; 168 HR post-dose on Cycle 1 Week 2; 504 HR post-dose) on Cycle 2 Week 1; Pre-dose on Week 1 of Cycles 4, 6, 12, 18, 24, 30, 36; End of Treatment (Up to approximately 196 weeks)
Population: PK population. The number analyzed for each timepoint reflects the number of participants from the Overall PK population with a non-missing value at the specified time point. Rows and Arms/Groups with 0 participants analyzed represent time points at which no participant data was available from within the respective Arms/Groups.
Measure: Mean (Standard Deviation); unit: milligram/ litre (mg/L)
Arm/Group | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 11 | 7 | 5 | 3
milligram/ litre (mg/L)
  Cycle 1 Week 1, Day 1 pre-dose | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Cycle 1 Week 1, 1 hr post-dose | 58.291 (10.7135) | 124.743 (30.9267) | 69.720 (9.8228) | 129.000 (2.6458)
  Cycle 1 Week 2, 168 hrs post-dose | 21.045 (4.5276) | 55.314 (10.1568) | 28.660 (14.1661) | 55.600 (8.2286)
  Cycle 2 Week 1, 504 hrs post-dose: number analyzed (Participants) | 9 | 6 | 3 | 2
  Cycle 2 Week 1, 504 hrs post-dose | 12.256 (2.1518) | 35.100 (11.1095) | 13.240 (5.0411) | 43.000 (7.4953)
  Cycle 4 Week 1, Pre-dose: number analyzed (Participants) | 1 | 1 | 0 | 0
  Cycle 4 Week 1, Pre-dose | 23.100 (NA) — Standard deviation is not evaluable as only single participant was analyzed. | 81.400 (NA) — Standard deviation is not evaluable as only single participant was analyzed. |  |
  Cycle 6 Week 1, Pre-dose: number analyzed (Participants) | 1 | 1 | 0 | 0
  Cycle 6 Week 1, Pre-dose | 25.100 (NA) — Standard deviation is not evaluable as only single participant was analyzed. | 103.000 (NA) — Standard deviation is not evaluable as only single participant was analyzed. |  |
  Cycle 12 Week 1, Pre-dose: number analyzed (Participants) | 1 | 1 | 0 | 0
  Cycle 12 Week 1, Pre-dose | 21.400 (NA) — Standard deviation is not evaluable as only single participant was analyzed. | 58.400 (NA) — Standard deviation is not evaluable as only single participant was analyzed. |  |
  Cycle 18 Week 1, Pre-dose: number analyzed (Participants) | 1 | 1 | 0 | 0
  Cycle 18 Week 1, Pre-dose | 21.200 (NA) — Standard deviation is not evaluable as only single participant was analyzed. | 60.900 (NA) — Standard deviation is not evaluable as only single participant was analyzed. |  |
  Cycle 24 Week 1, Pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 24 Week 1, Pre-dose | 12.400 (NA) — Standard deviation is not evaluable as only single participant was analyzed. |  |  |
  Cycle 30 Week 1, Pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 30 Week 1, Pre-dose | 33.800 (NA) — Standard deviation is not evaluable as only single participant was analyzed. |  |  |
  Cycle 36 Week 1, Pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 0
  Cycle 36 Week 1, Pre-dose | 33.500 (NA) — Standard deviation is not evaluable as only single participant was analyzed. |  |  |
  End of Treatment, End of Treatment: number analyzed (Participants) | 8 | 6 | 3 | 2
  End of Treatment, End of Treatment | 16.543 (8.6016) | 58.700 (47.2811) | 16.507 (13.6358) | 46.800 (40.5879)

13. Secondary Outcome: Part 1A and Part 1B: Number of Participants With Positive Anti-Drug Antibody (ADAs) to Dostarlimab
Description: Blood samples were collected for the analysis of the presence of ADAs using electrochemiluminescence. All samples were tested in screening and confirmatory assay, and positive samples were further characterized for antibody titers.
Time Frame: Up to approximately 196 weeks
Population: Immunogenicity (ADA) Population included all participants who received at least 1 dose of dostarlimab and who had at least 1 ADA sample with a result.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 11 | 7 | 5 | 3
Participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Part 1A and Part 1B: Number of Participants Answered Acceptability and Palatability of Niraparib Via Questionnaires
Description: The acceptability and palatability for participants who received niraparib tablet or TfOS were evaluated by using a questionnaire.
Time Frame: At Week 1 of Cycle 1
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 11 | 7 | 5 | 3
Participants | 11 | 7 | 5 | 2

15. Secondary Outcome: Part 2 Safety-run in: Objective Response Rate (ORR)
Description: ORR is the percentage of participants with a best overall response (BOR) of confirmed CR or PR, using RECIST v1.1 or INRC (neuroblastoma only) as determined by the Investigator. Per RECIST v1.1: CR is disappearance of all target lesions, with pathological lymph nodes <10 mm in short axis. PR is ≥30% decrease in sum of diameters of target lesions, referencing baseline sum (percent change from baseline). Per INRC: CR is resolution of all detectable disease, including soft tissue, bone, and bone marrow, with residual lesion measurements <10 mm and no tumor infiltration in the bone marrow or abnormal MIBG/FDG uptake. PR: Significant reduction in tumor burden, including a ≥30% decrease in primary or metastatic lesion size and ≥50% reduction in bone involvement (MIBG/FDG), with no new lesions and bone marrow infiltration ≤5%.
Time Frame: Up to approximately 196 weeks
Population: Intent-to-treat population included all participants who received any study medication and had measurable baseline tumour assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 3
Percentage of Participants | 0 [NA to NA] — No participants achieved confirmed CR or PR

16. Secondary Outcome: Part 2 Safety-run in: Duration of Response (DOR)
Description: DOR is the time from first documented response (CR or PR) to first PD by RECIST v1.1 or INRC (neuroblastoma only), based on Investigator assessment, or death (whichever occurs first). It is calculated for participants with a BOR of confirmed CR or PR. If no PD or death occurs post-response, participants are censored at their last tumor assessment date. Per RECIST v1.1, CR is disappearance of all target lesions; PR is ≥30% decrease in lesion diameters from baseline; PD is ≥20% increase in lesion sum from nadir plus ≥5 mm absolute increase. Per INRC, CR is resolution of detectable disease, including soft tissue, bone, and bone marrow, with residual lesions <10 mm, no bone marrow infiltration, and normal MIBG/FDG uptake. PR is a ≥30% decrease in lesion size, ≥50% reduction in bone involvement (MIBG/FDG), no new lesions, and bone marrow infiltration ≤5%. PD is >20% lesion size increase, new lesions, or increased infiltration in bone marrow.
Time Frame: Up to approximately 196 weeks
Population: ITT population. Only responders (CR or PR) by investigator assessment were included in this analysis.
Arm/Group | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 0

17. Secondary Outcome: Part 2 Safety-run in: Disease Control Rate (DCR)
Description: DCR is the percentage of participants achieving a BOR of confirmed CR, PR, or stable disease (SD) by RECIST v1.1 or INRC (neuroblastoma only). Per RECIST v1.1: CR is disappearance of all target lesions and pathological lymph nodes <10 mm in short axis; PR is ≥30% decrease in lesion diameters from baseline; SD is neither sufficient shrinkage for PR nor sufficient increase for PD. Per INRC: CR is resolution of all detectable disease (soft tissue, bone, marrow) with residual lesion <10 mm, no tumor infiltration in the bone marrow, and no abnormal MIBG or FDG/PET uptake. PR is ≥30% decrease in lesion size, ≥50% bone involvement reduction (MIBG/FDG uptake), no new lesions, and bone marrow infiltration ≤5%. SD was defined as neither sufficient shrinkage for PR nor sufficient increase for PD at the primary site. Bone marrow infiltration remains >5%.
Time Frame: Up to approximately 196 weeks
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 3
Percentage of Participants | 0 [NA to NA] — No participants with confirmed CR, PR or stable disease

18. Secondary Outcome: Part 2 Safety-run in: Progression-free Survival (PFS)
Description: PFS is defined as the time from the date of the first dose of study treatment to the first documented PD, as determined by RECIST v1.1 or INRC (in participants with neuroblastoma only) based on Investigator assessment, or death from any cause (whichever occurs first). Per RECISTv1.1: PD was defined as At least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm. Per INRC: PD is >20% lesion size increase, new lesions, or increased marrow tumor infiltration (>5%).
Time Frame: Up to approximately 196 weeks
Population: ITT population
Measure: Median (Full Range); unit: Months
Arm/Group | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 3
Months | 1.68 [1.35 to 2]

19. Secondary Outcome: Part 2 Safety-run in: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious AEs (SAEs)
Description: as for outcome 8
Time Frame: Up to approximately 196 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 3
Participants
  TEAEs | 3
  SAEs | 2

20. Secondary Outcome: Part 2 Safety-run in: Number of Participants With Dostarlimab-Related Immune-Mediated Adverse Events (imAEs)
Description: as for outcome 9
Time Frame: Up to approximately 196 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 3
Participants | 2

21. Secondary Outcome: Part 2 Safety-run in: Number of Participants With TEAEs Leading to Death and Treatment Discontinuation
Description: as for outcome 10
Time Frame: Up to approximately 196 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 3
Participants
  Leading to Death | 0
  Treatment Discontinuation | 2

22. Secondary Outcome: Part 2 Safety-run in: Niraparib Concentrations
Description: Blood samples were obtained to analyze niraparib concentration levels.
Time Frame: 2.5 HR and 7 HR post-dose on Cycle 1 Week 1, Pre-dose on Cycle 1 Week 2 and Pre-dose and 5 HR post-dose on Cycle 2 Week 1
Population: PK population. Only those participants with data available at specified data points have been analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg
Number analyzed (Participants) | 3
ng/mL
  Cycle 1 Week 1, 2.5 HR post-dose | 109.000 (121.7060)
  Cycle 1 Week 1, 7 HR post-dose | 292.067 (225.1404)
  Cycle 1 Week 2, Pre-dose | 329.200 (272.7140)
  Cycle 2 Week 1, Pre-dose | 338.667 (253.1291)
  Cycle 2 Week 1, 5 HR post-dose | 834.667 (612.8428)

23. Secondary Outcome: Part 2A: Objective Response Rate (ORR) by the Investigator Using RECIST v1.1
Description: ORR is defined as the percentage of participants who have a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) as determined by the Investigator using RECIST v1.1. CR was defined as disappearance of all target and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline).
Time Frame: Up to approximately 196 weeks
Population: Modified Intent-to-treat (mITT) population for Osteosarcoma cohort. Only those participants at specified timepoint have been anaysed. Data from 1 participant treated in Part 1A Cohort 1A at the same dose level as 8 participants treated in Part 2A were pooled and analyzed collectively for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma)
Number analyzed (Participants) | 9
Percentage of Participants | 0 [0.0 to 33.6]

24. Secondary Outcome: Part 2A: Duration of Response (DOR) by the Investigator Using RECIST v1.1
Description: DOR is defined as the time from first documentation of response (CR or PR) until the time of first documented PD by RECIST v1.1 , based on Investigator assessment, or death (whichever occurs first). CR was defined as disappearance of all target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline). PD was defined as At least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm.
Time Frame: Up to approximately 196 weeks
Population: Modified Intent-to-treat (mITT) population for Osteosarcoma cohort. Only responders (CR or PR) by investigator assessment were included in this analysis.
Arm/Group | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma)
Number analyzed (Participants) | 0

25. Secondary Outcome: Part 2A: Disease Control Rate (DCR) by the Investigator Using RECIST v1.1
Description: DCR is defined as the percentage of participants who have achieved a BOR of confirmed CR, confirmed PR, or stable disease (SD) by RECIST v1.1. CR was defined as disappearance of all target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline). SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Up to approximately 196 weeks
Population: Modified Intent-to-treat (mITT) population for Part 2A Osteosarcoma cohort. Data from 1 participant treated in Part 1A Cohort 1A at the same dose level as 8 participants treated in Part 2A were pooled and analyzed collectively for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma)
Number analyzed (Participants) | 9
Percentage of Participants | 0 [0.0 to 33.6]

26. Secondary Outcome: Part 2A: Progression-free Survival (PFS) by the Investigator Using RECIST v1.1
Description: PFS is defined as the time from the date of the first dose of study treatment to the first documented PD, as determined by RECIST v1.1 , based on Investigator assessment, or death from any cause (whichever occurs first). PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start).
Time Frame: Up to approximately 196 weeks
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma)
Number analyzed (Participants) | 9
Months | 1.2 [0.7 to 2.1]

27. Secondary Outcome: Part 2A: Number of Participants With of Treatment Emergent Adverse Events (TEAEs) and Serious AEs (SAEs)
Description: as for outcome 8
Time Frame: Up to approximately 196 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma)
Number analyzed (Participants) | 11
Participants
  TEAEs | 11
  SAEs | 4

28. Secondary Outcome: Part 2A: Number of Participants With Dostarlimab-Related Immune-Mediated Adverse Events (imAEs)
Description: as for outcome 9
Time Frame: Up to approximately 196 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma)
Number analyzed (Participants) | 11
Participants | 2

29. Secondary Outcome: Part 2A: Number of Participants With TEAEs Leading to Death and Treatment Discontinuation
Description: as for outcome 10
Time Frame: Up to approximately 196 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma)
Number analyzed (Participants) | 11
Participants
  Leading to Death | 0
  Treatment Discontinuation | 2

30. Secondary Outcome: Part 2A: Niraparib Concentrations
Description: Blood samples were obtained to analyze niraparib concentration levels.
Time Frame: 2.5 HR and 7 HR post-dose on Cycle 1 Week 1, 168 HR post-dose on Cycle 1 Week 2
Population: PK population. Only those participants with data available at specified data points have been analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma)
Number analyzed (Participants) | 11
ng/mL
  Cycle 1 Week 1, 2.5 HR post-dose | 217.212 (236.5667)
  Cycle 1 Week 1, 7 HR post-dose | 241.482 (143.3515)
  Cycle 1 Week 2, 168 HR post-dose: number analyzed (Participants) | 10
  Cycle 1 Week 2, 168 HR post-dose | 354.100 (153.7909)

31. Secondary Outcome: Part 2A: Dostarlimab Concentrations
Description: Blood samples were collected for PK analysis of Dostarlimab.
Time Frame: Pre-dose on Day 1; 1 HR post-dose on Cycle 1 Week 1; 168 HR post-dose on Cycle 1 Week 2; 504 HR post-dose) on Cycle 2 Week 1; Pre-dose on Week 1 of Cycles 4 and 6; End of Treatment (Up to approximately 196 weeks)
Population: PK population. Only those participants with data available at specified data points have been analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma)
Number analyzed (Participants) | 11
mg/L
  Cycle 1 Week 1, Day 1 pre-dose | 0.000 (0.0000)
  Cycle 1 Week 1, 1 hr post-dose | 135.509 (45.2007)
  Cycle 1 Week 2, 168 hrs post-dose: number analyzed (Participants) | 9
  Cycle 1 Week 2, 168 hrs post-dose | 65.022 (8.6129)
  Cycle 2 Week 1, 504 hrs post-dose: number analyzed (Participants) | 9
  Cycle 2 Week 1, 504 hrs post-dose | 45.000 (27.4571)
  Cycle 4 Week 1, Pre-dose: number analyzed (Participants) | 2
  Cycle 4 Week 1, Pre-dose | 46.900 (23.0517)
  Cycle 6 Week 1, Pre-dose: number analyzed (Participants) | 1
  Cycle 6 Week 1, Pre-dose | 133.000 (NA) — Standard deviation is not evaluable as only single participant was analyzed.
  End of Treatment, End of Treatment: number analyzed (Participants) | 8
  End of Treatment, End of Treatment | 74.338 (52.2281)

32. Secondary Outcome: Part 2A: Number of Participants With Positive Anti-Drug Antibody (ADAs) to Dostarlimab
Description: as for outcome 13
Time Frame: Up to approximately 196 weeks
Population: ADA Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma)
Number analyzed (Participants) | 10
Participants | 0

33. Secondary Outcome: Part 2A: Number of Participants Answered Acceptability and Palatability of Niraparib Via Questionnaires
Description: The acceptability and palatability for participants who received niraparib tablet were evaluated by using a questionnaire.
Time Frame: At Week 1 of Cycle 1
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma)
Number analyzed (Participants) | 11
Participants | 11

34. Secondary Outcome: Part 2B: Duration of Response (DOR) by the Investigator by INRC
Description: DOR is defined as the time from first documentation of response (CR or PR) until the time of first documented PD by INRC , based on Investigator assessment, or death (whichever occurs first). CR is resolution of all detectable disease, including soft tissue, bone, and bone marrow, with residual lesion measurements <10 mm and no tumor infiltration in the bone marrow or abnormal MIBG/FDG uptake. PR: Significant reduction in tumor burden, including a ≥30% decrease in primary or metastatic lesion size and ≥50% reduction in bone involvement (MIBG/FDG), with no new lesions and bone marrow infiltration ≤5%. PD is >20% lesion size increase,new lesions or increased tumor infiltration in bone marrow.
Time Frame: Up to approximately 196 weeks
Population: Modified Intent-to-treat (mITT) population for Part 2B Neuroblastoma cohort. Only responders (CR or PR) by investigator assessment were included in this analysis.
Arm/Group | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma)
Number analyzed (Participants) | 0

35. Secondary Outcome: Part 2B: Disease Control Rate (DCR) by the Investigator by INRC
Description: DCR is defined as the percentage of participants who have achieved a BOR of confirmed CR, confirmed PR, or SD by INRC. CR is resolution of all detectable disease (soft tissue, bone, marrow) with residual lesion <10 mm, no tumor infiltration in the bone marrow, and no abnormal MIBG or FDG/PET uptake. PR is ≥30% decrease in lesion size, ≥50% bone involvement reduction (MIBG/FDG uptake), no new lesions, and bone marrow infiltration ≤5%. SD was defined as neither sufficient shrinkage for PR nor sufficient increase for PD at the primary site. Bone marrow infiltration remains >5%.
Time Frame: Up to approximately 196 weeks
Population: Modified Intent-to-treat (mITT) population for Part 2B Neuroblastoma cohort. Data from 2 participants treated in Part 1A Cohort 1A at the same dose level as 6 participants treated in Part 2B were pooled and analyzed collectively for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma)
Number analyzed (Participants) | 8
Percentage of Participants | 38 [8.5 to 75.5]

36. Secondary Outcome: Part 2B: Progression-free Survival (PFS) by the Investigator by INRC
Description: PFS is defined as the time from the date of the first dose of study treatment to the first documented PD, as determined by INRC , based on Investigator assessment, or death (whichever occurs first). PD is >20% lesion size increase, new lesions, or increased tumor infiltration in bone marrow.
Time Frame: Up to approximately 196 weeks
Population: as for outcome 35
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma)
Number analyzed (Participants) | 8
Months | 2.9 [0.5 to 10.2]

37. Secondary Outcome: Part 2B: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious AEs (SAEs)
Description: as for outcome 8
Time Frame: Up to approximately 196 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma)
Number analyzed (Participants) | 7
Participants
  TEAEs | 7
  SAEs | 4

38. Secondary Outcome: Part 2B: Number of Participants With Dostarlimab-Related Immune-Mediated Adverse Events (imAEs)
Description: as for outcome 9
Time Frame: Up to approximately 196 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma)
Number analyzed (Participants) | 7
Participants | 4

39. Secondary Outcome: Part 2B: Number of Participants With TEAEs Leading to Death and Treatment Discontinuation
Description: A TEAE is any event that emerged during treatment and was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment.
Time Frame: Up to approximately 196 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma)
Number analyzed (Participants) | 7
Participants
  Leading to Death | 0
  Treatment Discontinuation | 3

40. Secondary Outcome: Part 2B: Niraparib Concentrations
Description: Blood samples were obtained to analyze niraparib concentration levels.
Time Frame: 2.5 HR and 7 HR post-dose on Cycle 1 Week 1, 168 HR post-dose on Cycle 1 Week 2
Population: PK population. Only those participants with data available at specified data points have been analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma)
Number analyzed (Participants) | 7
ng/mL
  Cycle 1 Week 1, 2.5 HR post-dose | 275.600 (330.9424)
  Cycle 1 Week 1, 7 HR post-dose | 329.571 (182.8432)
  Cycle 1 Week 2, 168 HR post-dose | 700.143 (571.6900)

41. Secondary Outcome: Part 2B: Dostarlimab Concentrations
Description: Blood samples were collected for PK analysis of Dostarlimab.
Time Frame: Pre-dose on Day 1; 1 HR post-dose on Cycle 1 Week 1; 168 HR post-dose on Cycle 1 Week 2; 504 HR post-dose on Cycle 2 Week 1; Pre-dose on Week 1 of Cycles 4, 6, 12 and 18; End of Treatment (Up to approximately 196 weeks)
Population: PK population. Only those participants with data available at specified data points have been analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma)
Number analyzed (Participants) | 7
mg/L
  Cycle 1 Week 1, Day 1 pre-dose | 0.000 (0.0000)
  Cycle 1 Week 1, 1 hr post-dose | 186.000 (117.4748)
  Cycle 1 Week 2, 168 hrs post-dose | 61.943 (13.5405)
  Cycle 2 Week 1, 504 hrs post-dose: number analyzed (Participants) | 4
  Cycle 2 Week 1, 504 hrs post-dose | 39.925 (13.4205)
  Cycle 4 Week 1, Pre-dose: number analyzed (Participants) | 3
  Cycle 4 Week 1, Pre-dose | 88.500 (22.3900)
  Cycle 6 Week 1, Pre-dose: number analyzed (Participants) | 3
  Cycle 6 Week 1, Pre-dose | 173.667 (90.4231)
  Cycle 12 Week 1, Pre-dose: number analyzed (Participants) | 2
  Cycle 12 Week 1, Pre-dose | 179.500 (24.7487)
  Cycle 18 Week 1, Pre-dose: number analyzed (Participants) | 1
  Cycle 18 Week 1, Pre-dose | 121.000 (NA) — Standard deviation is not evaluable as only single participant was analyzed.
  End of Treatment, End of Treatment: number analyzed (Participants) | 5
  End of Treatment, End of Treatment | 93.580 (69.6794)

42. Secondary Outcome: Part 2B: Number of Participants With Positive Anti-Drug Antibody (ADAs) to Dostarlimab
Description: as for outcome 13
Time Frame: Up to approximately 196 weeks
Population: ADA Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma)
Number analyzed (Participants) | 7
Participants | 0

43. Secondary Outcome: Part 2B: Number of Participants Answered Acceptability and Palatability of Niraparib Via Questionnaires
Description: as for outcome 33
Time Frame: At Week 1 of Cycle 1
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma)
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: All cause mortality, non-SAEs and SAEs were collected upto approximately 196 weeks.
Description: The Safety Population included all participants who received at least 1 dose of either niraparib or dostarlimab.
Arm/Group | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma) | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma) | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg
All-Cause Mortality (participants affected / at risk) | 7/11 | 3/7 | 3/5 | 3/3 | 2/11 | 2/7 | 1/3
Serious Adverse Events (participants affected / at risk) | 6/11 | 2/7 | 2/5 | 2/3 | 4/11 | 4/7 | 2/3
Other Adverse Events (participants affected / at risk) | 11/11 | 7/7 | 5/5 | 3/3 | 11/11 | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) (N=11) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (N=7) | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg (N=5) | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg (N=3) | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma) (N=11) | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma) (N=7) | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated encephalitis (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A Cohort 0: Niraparib 100 Milligram (mg) + Dostarlimab 3 mg/Kilogram (kg) (N=11) | Part 1A Cohort 1A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (N=7) | Part 1A Cohort 1B: Niraparib 200 mg + Dostarlimab 3 mg/kg (N=5) | Part 1B Cohort 1: Niraparib AAOLF (Age-based Dose) + Dostarlimab 7.5 mg/kg (N=3) | Part 2A: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Osteosarcoma) (N=11) | Part 2B: Niraparib 100 mg + Dostarlimab 7.5 mg/kg (Neuroblastoma) (N=7) | Part 2: Safety- Run-In Niraparib TfOS (Weight-based Dose) + Dostarlimab 7.5 mg/kg (N=3)
Anaemia (Blood and lymphatic system disorders) | 7 (12) | 3 (5) | 2 (8) | 3 (6) | 3 (9) | 3 (8) | 2 (3)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 2 (4) | 0 (0) | 2 (3) | 0 (0) | 3 (8)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 2 (6) | 1 (4) | 1 (5) | 3 (9) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (4) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (4) | 3 (3) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (5) | 3 (4) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 4 (7) | 2 (3) | 1 (3) | 3 (3) | 3 (4) | 0 (0)
Asthenia (General disorders) | 3 (7) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 7 (13) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatosplenomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes dermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (5) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (3)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (5) | 1 (1) | 2 (3) | 1 (1) | 3 (5) | 1 (3)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 1 (4) | 1 (1) | 1 (2) | 0 (0)
Blood fibrinogen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (3) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Lipase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 2 (5) | 0 (0) | 1 (5) | 3 (7) | 0 (0)
Platelet count decreased (Investigations) | 2 (5) | 1 (1) | 1 (2) | 2 (8) | 1 (1) | 2 (5) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tri-iodothyronine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (5) | 2 (4) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (5) | 2 (5) | 0 (0) | 1 (3) | 2 (2) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT04544995/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT04544995/SAP_001.pdf